CLINICAL TRIAL: NCT01612845
Title: Platelet-Rich Fibrin for Arthroscopically Repaired Massive Rotator Cuff Tears: A Prospective Randomized Pilot Clinical Trial
Brief Title: Effect of Platelet-rich Fibrin on Rotator Cuff Repair
Acronym: PRP-Fibrin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: spanish society of orthopedics and traumatology (Unknown)
Responsible Party: Principal Investigator, Samuel Antuna, Consultant in Shoulder and Elbow Surgery, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-523
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Rotator Cuff Tears of the Shoulder
Keywords: rotator cuff; shoulder; platelet rich plasma; fibrin
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRF (Experimental): the group in which the PRF was administered
  Interventions: Biological: PRF (vivostat ®) administration after rotator cuff repair
- Control (Active Comparator): repair without PRF
  Interventions: Procedure: Arthroscopic repair without platelet rich fibrin

INTERVENTIONS:
Procedure: Arthroscopic repair without platelet rich fibrin — after the tendon is repaired, no additional procedures are performed and no PRF is administered
  Arms: Control
Biological: PRF (vivostat ®) administration after rotator cuff repair — 7cc. of autologous PRF are locally administered to the repair site after reconstruction of the rotator cuff
  Arms: PRF

SUMMARY:
The objective of this study was to prospectively evaluate the influence of local application of Platelet Rich Fibrin (PRF) on the functional outcome and integrity of the arthroscopically repaired tendons in patients with massive tears of the rotator cuff.

DETAILED DESCRIPTION:
A prospective, randomized clinical trial was performed on 28 patients (22 females, 6 males) with an average age of 65 years (range, 53 to 77) undergoing complete arthroscopic repair of a massive rotator cuff tear. In 14 patients, after the repair was completed, 6 cc. of PRF (vivostat ®) were locally applied to the repair site. In 14 patients no addition of PRF was performed. All patients underwent an arthro-MRI to evaluate the integrity of the repair and a clinical exam one year after the operation. All patients were then followed clinically at a minimum of 2 years. Functional outcome was evaluated with the Constant and DASH scores.

ELIGIBILITY:
Inclusion Criteria:

* Massive rotator cuff tears affecting supraspinatus and infraspinatus
* Failed conservative treatment for at least 6 months
* No hematologic disorder

Exclusion Criteria:

* Rotator cuff affecting subscapularis
* chronic infectious disease
* anemia
* clot disorders
* low platelet count
* history of difficulty in venous puncture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
rotator cuff tear healing rate after surgical reconstruction evaluated by arthro-MRI | one year

SECONDARY OUTCOMES:
functional outcome evaluated with constant score | two years
disability outcome evaluated with dash score | two years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Antuña, MD PhD, Study Director — H. La PAz; Raul Barco, MD PhD, Principal Investigator — HU La PAz; Jose M Martinez, MD, Principal Investigator — HU La Paz; Jose M sanchez, MD, Principal Investigator — HU La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Jo CH, Kim JE, Yoon KS, Lee JH, Kang SB, Lee JH, Han HS, Rhee SH, Shin S. Does platelet-rich plasma accelerate recovery after rotator cuff repair? A prospective cohort study. Am J Sports Med. 2011 Oct;39(10):2082-90. doi: 10.1177/0363546511413454. Epub 2011 Jul 7. PMID 21737832
- [Background] Randelli P, Arrigoni P, Ragone V, Aliprandi A, Cabitza P. Platelet rich plasma in arthroscopic rotator cuff repair: a prospective RCT study, 2-year follow-up. J Shoulder Elbow Surg. 2011 Jun;20(4):518-28. doi: 10.1016/j.jse.2011.02.008. PMID 21570659
- [Background] Castricini R, Longo UG, De Benedetto M, Panfoli N, Pirani P, Zini R, Maffulli N, Denaro V. Platelet-rich plasma augmentation for arthroscopic rotator cuff repair: a randomized controlled trial. Am J Sports Med. 2011 Feb;39(2):258-65. doi: 10.1177/0363546510390780. Epub 2010 Dec 15. PMID 21160018
- [Result] Barber FA, Hrnack SA, Snyder SJ, Hapa O. Rotator cuff repair healing influenced by platelet-rich plasma construct augmentation. Arthroscopy. 2011 Aug;27(8):1029-35. doi: 10.1016/j.arthro.2011.06.010. PMID 21802625